CLINICAL TRIAL: NCT02887417
Title: Glioblastoma Platelet Activation Study
Acronym: GPAS
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Sascha Marx, Dr. med., University Medicine Greifswald
Other Study IDs: Glioma-HGW
Record Dates: First submitted 2016-08-18; First posted 2016-09-02 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Glioblastoma; Circulating Platelet-monocyte Conjugates
Keywords: platelet activation
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients: glioblastoma patients
- controls: healthy controls

SUMMARY:
Glioblastoma face an increased risk of venous or arterial thromboembolism. Furthermore, the most frequent immune cells in glioblastoma are tumor associated macrophages, which find theirself in an anti-inflammatory (M2) phenotype.

Increased conjugates between circulating platelets and monocytes reflect an pro-inflammatory status.

DETAILED DESCRIPTION:
Glioblastoma face an increased risk of venous or arterial thromboembolism. Furthermore, the most frequent immune cells in glioblastoma are tumor associated macrophages, which find theirself in an anti-inflammatory (M2) phenotype.

Increased conjugates between circulating platelets and monocytes reflect an pro-inflammatory status.

ELIGIBILITY:
Inclusion Criteria:

* MR-morphological suspicion for glioblastoma
* informed consent

Exclusion Criteria:

* no informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consecutive patients with suspicious for glioblastoma
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mean P-selectine expression in all platelets | 01/ 2016 - 10/ 2016
Mean CD63 expression in all platelets | 01/ 2016 - 10/ 2016
Mean CD40 Expression in all platelets | 01/ 2016 - 10/ 2016
Mean platelet-monocyte-conjugate formation in the monocyte population | 01/ 2016 - 10/ 2016

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Greifswald, Germany